CLINICAL TRIAL: NCT05412173
Title: A Randomized, Open-label, Cross-over Adaptive Study of the Comparative Pharmacokinetics and Bioequivalence of the Drugs Molnupiravir, Capsules, 200 mg and Lagevrio, Capsules, 200 mg in Healthy Volunteers at Fasted Conditions
Brief Title: Pharmacokinetics and Bioequivalence of Molnupiravir, 200 mg Capsules and Lagevrio, 200 mg Capsules in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MOL-05-02-2021
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Viral Infection; COVID-19
MeSH Terms: conditions — Virus Diseases; COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT-sequence (Other): The volunteers will take 1 capsule (200 mg) of Lagevrio (R), 200 mg capsules (Merck Sharp & Dohme (UK) Limited, UK) in Period 1, and 1 capsule (200 mg) of Molnupiravir (T), 200 mg capsules (Valenta Pharm, Russia) in Period 2.
  Interventions: Drug: Molnupiravir
- TR-sequence (Other): The volunteers will take 1 capsule (200 mg) of the drug Molnupiravir (T), capsules, 200 mg (Valenta Pharm JSC, Russia) in Period 1, and 1 capsule (200 mg) of the drug Lagevrio (R), capsules, 200 mg (Merck Sharp & Dohme (UK) Limited, UK) in Period 2.
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Molnupiravir — A single dose of R or T drug in each of 2 periods of the study in fasted conditions

SUMMARY:
The study aimed for:

1. Comparative evaluation of the safety of the drug Molnupiravir, capsules, 200 mg (JSC "Valenta Pharm", Russia), and Lagevrio, capsules, 200 mg (Merck Sharp & Dohme (UK) Limited, UK), based on the analysis of adverse events (AEs);
2. Comparative assessment of pharmacokinetic parameters and bioequivalence of the drug Molnupiravir, capsules, 200 mg (Valenta Pharm JSC, Russia), and Lagevrio, capsules, 200 mg (Merck Sharp & Dohme (UK) Limited, UK), in healthy volunteers in fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of written consent of the volunteer to participate in the study in accordance with applicable law.
2. Healthy male and female caucasian volunteers aged 18 to 45 years (inclusive).
3. Verified diagnosis "healthy": no deviations from the reference values of the data of standard clinical, laboratory and instrumental methods of examination.
4. Systolic blood pressure (SBP) in the range of 110-130 mmHg; diastolic blood pressure (DBP) is 60-85 mmHg).
5. 60-90 bpm at rest for heart rate (HR).
6. 16-20 breaths/min for respiratory rate (RR).
7. 35.5 to 36.9°C for body temperature.
8. Body mass index (BMI) within the range of 18.5 ≤ BMI ≤ 30 kg/m2 with a body weight not less than 45 kg for female and not less than 55 kg for male volunteers.
9. The consent of the volunteer (including the partner) to use adequate methods of contraception during the study and 30 days after its completion; for female volunteers - negative blood/urine test result for β-chorionic gonadotropin.
10. Volunteers must behave adequately, coherent speech must be observed.

Exclusion Criteria:

1. A history of allergy;
2. A history of drug intolerance to the active and/or excipients in the study drugs;
3. Chronic diseases of the kidneys, liver, gastrointestinal tract (GIT), cardiovascular, lymphatic, respiratory, nervous, endocrine, musculoskeletal, genitourinary and immune systems, as well as skin, blood and vision;
4. History of gastrointestinal surgery (except appendectomy at least 1 year prior to screening);
5. Diseases/conditions that in the opinion of the investigator may affect the absorption, distribution, metabolism or excretion of the study drugs (drugs);
6. Acute infectious disease less than 4 weeks prior to screening;
7. Taking medications that significantly affect hemodynamics and medications that affect liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months prior to screening;
8. Regularly taking a medicines less than 2 weeks before screening and taking a single medicine less than 7 days before screening;
9. Donating blood or plasma less than 3 months before screening;
10. Use of hormonal contraceptives (in women) less than 2 months before screening;
11. The use of depot injections of any drug less than 3 months before screening;
12. Pregnancy or lactation; positive blood/urine β-CGH test for women with preserved reproductive potential;
13. Women of preserved reproductive potential with a history of unprotected intercourse within 30 days prior to study drug administration with an unsterilized partner;
14. Participation in another clinical trial less than 3 months prior to screening or concurrently with the present study;
15. Taking more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 mL of beer, 150 mL of wine or 40 mL of spirits) in the week in the last month before inclusion in the study or anamnestic evidence of alcoholism, drug addiction, drug abuse;
16. Smoking more than 10 cigarettes per day currently, or a history of smoking the specified number of cigarettes during the 6 months prior to screening; disagreement to abstain from smoking for the duration of the hospital stay;
17. Positive blood tests for antibodies to human immunodeficiency virus (HIV) 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens, rapid tests of biomaterial (nasopharyngeal and/or oropharyngeal swab) for Severe Acute Respiratory Syndrome Coronavirus 2 antigen (SARS-CoV-2), Coronavirus Disease 2019 (COVID-19);
18. Clinically significant abnormalities on the electrocardiogram (ECG);
19. Positive urinalysis for narcotics and potent drugs;
20. Positive test for the content of alcohol vapor in exhaled air.
21. Scheduling an inpatient stay during the study period, for any reason other than hospitalization required by this protocol.
22. Inability to meet the requirements of the protocol, perform the procedures prescribed in the protocol, follow the diet, activity regimen.
23. Other conditions that, in the opinion of the Investigator, preclude inclusion of the volunteer in the study or may result in early withdrawal of the volunteer from the study, including fasting or a special diet (e.g. vegetarian, vegan, limited table salt) or a special lifestyle (night work, extreme physical activity).

Withdrawal criteria:

1. A volunteer withdraws from further participation in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Occurrence of causes/occurrence during the study of situations that threaten the safety of the volunteer (e.g., hypersensitivity reactions, etc.);
4. Volunteers selected for the study in violation of the inclusion/inclusion criteria;
5. Volunteer's development of severe adverse event during the study;
6. Missing 2 or more consecutive blood samples or 3 or more blood samples during the same Study Period.
7. Occurrence of vomiting/diarrhea within 6 hours of study drug administration;
8. Positive urine test for narcotics and drugs;
9. Positive breath alcohol vapor test.
10. Positive pregnancy test in women;
11. Positive test for COVID-19;
12. The occurrence in the course of the study of other reasons that prevent the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Maximum plasma concentration (Cmax) of β-D-N-4-hydroxycytidine (NHC)
Pharmacokinetics - tmax | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Time to reach Cmax (tmax) of NHC
Pharmacokinetics - AUC0-t | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of NHC
Pharmacokinetics - AUC0-inf | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of NHC
Pharmacokinetics - AUCextr | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Extrapolated AUC of NHC, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Elimination half-life (t1/2) of NHC
Pharmacokinetics - kel | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Elimination constant (kel) of NHC
Pharmacokinetics - MRT | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Mean residence time (MRT) of NHC
Bioequivalence - ratio of Cmax | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean Cmax for NHC after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-t | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean AUC0-t for NHC after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-inf | From 0 to 24 hours (Day 1-2 and Day 8-9)
  Ratio of geometric mean AUC0-inf for NHC after intake of R or T (with 90% confidence intervals)

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 14 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 14)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: adverse event (AE) characteristics | From the screening (and signing informed consent form) to Day 14 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 14)
  Description and severity of AEs or serious AEs (SAEs), concomitant therapy for AEs/SAEs, causal relationship, outcomes.
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Physical examination results
Safety and Tolerability: urinalysis - color | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  pH of the urine
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - nitrites | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Nitrites in the urine (+/-)
Safety and Tolerability: urinalysis - protein | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis - ketones | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Ketones in the urine (mmol/L)
Safety and Tolerability: urinalysis - urobilinogen | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Urobilinogen in the urine (mmol/L)
Safety and Tolerability: urinalysis - bilirubin | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Bilirubin in the urine (+/-)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders (except hyaline) | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Cylinders (except hyaline) in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Bacteria in the urine (number in sight)
Safety and Tolerability: complete blood count - hemoglobin | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - neutrophils | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Neutrophils, %
Safety and Tolerability: complete blood count - lymphocytes | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Basophils, %
Safety and Tolerability: blood test results - total protein | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - urea | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Urea in blood serum, mmol/L
Safety and Tolerability: blood test results - glucose | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - direct bilirubin | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Direct bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - triglycerides | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  Triglycerides in blood serum, mmol/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  ALP in blood serum, U/L
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening, Day 3, Day 9 or on early termination visit within the time frame of the study (from Day 0 to Day 14)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "Research Center Eco-Safety", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided